CLINICAL TRIAL: NCT02775877
Title: Letrozole and Sequential Clomiphene to Improve the Outcome of Embryo Transfer in Polycystic Ovary Syndrome (PCOS) Patients
Brief Title: Letrozole and Sequential Clomiphene to Improve the Outcome of Embryo Transfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Yunhai Chuai, Department of Obstetrics and Gynecology, Navy General Hospital, Beijing, Navy General Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HL2015
Record Dates: First submitted 2015-12-29; First posted 2016-05-18 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Female Infertility Due to Nonimplantation of Ovum
Keywords: PCOS; letrozole; clomiphene
MeSH Terms: interventions — Letrozole; Clomiphene

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- letrozole and clomiphene (Experimental): Letrozole 5 mg tablet orally from 3-7 day of once a day menstrual cycle and clomiphene100 mg tablet orally once a day from 11-15 day of menstrual cycle.
  Interventions: Drug: Letrozole; Drug: clomiphene
- Letrozole and human menopausal gonadotropin (HMG) (Active Comparator): Letrozole 5 mg tablet orally from 3-7 day of once a day menstrual cycle and HMG 75u once a day by intramuscular injection from 11-15day of menstrual cycle
  Interventions: Drug: Letrozole; Drug: HMG

INTERVENTIONS:
Drug: Letrozole
Drug: clomiphene
  Arms: letrozole and clomiphene
Drug: HMG
  Arms: Letrozole and human menopausal gonadotropin (HMG)

SUMMARY:
The purpose of this study is to study the effects of letrozole and sequential clomiphene in ovulation and pregnancy in PCOS patients.

DETAILED DESCRIPTION:
To evaluate the efficacy of letrozole and clomiphene in PCOS patients is important,especially in resistent PCOS patients. Although most medications prove the effectiveness of letrozole and clomiphene,the subjects of letrozole and sequential clomiphene in PCOS patients are rarely.The trial may provide further basis for this medication in PCOS patients in ovulation. If the medication demonstrates efficacy, the method would help the patients with PCOS to deal with the problem of infertility.

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS

Exclusion Criteria:

* •Women more than 38 years or less than 20 years

  * With infectious diseases or endocrine diseases
  * Who refuse to participate in the experiment

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-06 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
live birth rate | 3 years
  The event that a FETUS is born alive with heartbeats or RESPIRATION

SECONDARY OUTCOMES:
clinical pregnancy rate | 3 years
  The ratio of the number of conceptions (CONCEPTION) including Live BIRTH; STILLBIRTH; and fetal losses, to the mean number of females of reproductive age in a population during a set time period.
multiple pregnancies | 3 years
  The condition of carrying two or more FETUSES.
miscarriage | 3 years
  Expulsion of the product of FERTILIZATION before completing the term of GESTATION and without deliberate interference.
mature follic | 1 month
  The diameter of follic more than 18mm is the mature follic

CONTACTS AND LOCATIONS:
Overall Officials: Aiming Wang, Dr, Principal Investigator — Navy General Hospital, Beijing
Locations (1):
- Department of Obstetrics and Gynecology, Navy General Hospital., Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kamath MS, George K. Letrozole or clomiphene citrate as first line for anovulatory infertility: a debate. Reprod Biol Endocrinol. 2011 Jun 21;9:86. doi: 10.1186/1477-7827-9-86. PMID 21693034
- [Background] Legro RS, Kunselman AR, Brzyski RG, Casson PR, Diamond MP, Schlaff WD, Christman GM, Coutifaris C, Taylor HS, Eisenberg E, Santoro N, Zhang H; NICHD Reproductive Medicine Network. The Pregnancy in Polycystic Ovary Syndrome II (PPCOS II) trial: rationale and design of a double-blind randomized trial of clomiphene citrate and letrozole for the treatment of infertility in women with polycystic ovary syndrome. Contemp Clin Trials. 2012 May;33(3):470-81. doi: 10.1016/j.cct.2011.12.005. Epub 2012 Jan 13. PMID 22265923
- [Result] Hajishafiha M, Dehghan M, Kiarang N, Sadegh-Asadi N, Shayegh SN, Ghasemi-Rad M. Combined letrozole and clomiphene versus letrozole and clomiphene alone in infertile patients with polycystic ovary syndrome. Drug Des Devel Ther. 2013 Dec 3;7:1427-31. doi: 10.2147/DDDT.S50972. eCollection 2013. PMID 24348019
- [Result] Legro RS, Zhang H; Eunice Kennedy Shriver NICHD Reproductive Medicine Network. Letrozole or clomiphene for infertility in the polycystic ovary syndrome. N Engl J Med. 2014 Oct 9;371(15):1463-4. doi: 10.1056/NEJMc1409550. No abstract available. PMID 25295506